CLINICAL TRIAL: NCT07240363
Title: First Line Surgery or First Line Fertility Treatment Using Assisted Reproductive Technologies in Patients With Advanced Endometriosis: A National Multicenter Randomized-controlled Trial
Brief Title: First Line Surgery or First Line Fertility Treatment Using Assisted Reproductive Technologies in Patients With Advanced Endometriosis
Acronym: EndoSOFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); The Swedish Medical Association (Other); Forte (Industry); Västra Götalandsregionen (Other)
Responsible Party: Principal Investigator, Malin Brunes, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-04293-01
Record Dates: First submitted 2025-10-02; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis; Infertility Assisted Reproductive Technology
Keywords: Endometriosis; Infertility; Surgery; ART
MeSH Terms: conditions — Endometriosis; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First-line ART (No Intervention): Women allocated in the ART arm will undergo up to three cycles of controlled ovarian stimulation (COS) followed by oocyte retrievals and embryo transfers. In Sweden, ART-treatment costs for women under the age of forty and without having children in current relationship are covered by the tax-funded healthcare system, with up to 3 IVF/ICSI treatments, given that they are considered medically meaningful, and that each stimulation is started before the woman turns 40 years of age (39). In case the treatment results in cryopreserved embryos, it is planned that they should be transferred prior to the start of any new COS. Women will be managed according to a routine clinical protocol at each reproductive unit. Stimulation protocols will be chosen individually by clinicians, taking into consideration age and ovarian reserve of each woman, as it is a standard routine in the collaborating Reproductive Units.
- First-line surgery followed by ART (Experimental): Surgery will be performed at one of four nationally specialized centers in advanced endometriosis surgery (Södersjukhuset Stockholm, Sahlgrenska University Hospital Göteborg, Skånes University Hospital, Malmö/Lund, Uppsala University Hospital). Surgery will be conducted according to the ESHRE recommendations of surgery in endometriomas and deep endometriosis (32, 33). Surgery should be multidisciplinary when needed (colorectal surgeons and urologists). The goal of the procedure is to remove as many endometriotic lesions as possible while also minimizing negative impact on organ function, since endometriosis is a benign disease. Rectal endometriosis will be removed with rectal shaving, discoid or segmental resection depending on the size and placement of the lesion in the rectal wall. Laparoscopic cyst enucleation is considered the "golden standard". In cases where ovarian reserve is already diminished, more gentle ablation methods could be employed
  Interventions: Procedure: Endometriosis surgery

INTERVENTIONS:
Procedure: Endometriosis surgery — Endometriosis surgery followed by ART
  Arms: First-line surgery followed by ART

SUMMARY:
Endometriosis is a chronic disease affecting approximately 10% of women of reproductive age. It is strongly associated with pelvic pain and infertility. Women with advanced stages of the disease (stage III-IV) have markedly reduced fertility compared with the general population. A Swedish study has shown that about 22% of women undergoing treatments with assisted reproductive technologies (ART), such as in vitro fertilization (IVF), are affected by endometriosis.

The optimal management of women with advanced endometriosis and infertility remains uncertain. Some clinicians advocate proceeding directly to IVF, while others suggest surgical removal of endometriosis lesions prior to IVF in order to improve the chances of pregnancy. Currently, evidence is limited to a small number of observational studies. Two observational studies and one meta-analysis have suggested that surgery before IVF in women with deep endometriosis may increase both pregnancy and live birth rates compared with IVF alone. However, no randomized controlled trial (RCT) has yet been conducted to answer this important clinical question.

This study will be the first national multicenter randomized controlled trial to compare surgery followed by IVF with IVF alone in women with advanced endometriosis and infertility. All Swedish centers for highly specialized endometriosis surgery and fertility treatment will participate.

Eligible participants are women under 39 years of age with stage III-IV endometriosis who seek fertility treatment. Participants will be randomized in a 1:1 ratio to one of two groups:

* Surgery prior to IVF (laparoscopic excision of endometriosis lesions, followed by IVF).
* Direct IVF without prior surgery. The primary outcome is the cumulative live birth rate within three years of randomization and initiation of the allocated treatment. Secondary outcomes include pregnancy rates, time to pregnancy, treatment-related complications, patient-reported quality of life, and cost-effectiveness.

Our hypothesis is that surgery before IVF will lead to a higher cumulative live birth rate compared with IVF without prior surgery in women with advanced endometriosis.

The results of this trial are expected to have significant impact on clinical practice and international guidelines. Regardless of outcome, the study will provide robust evidence to guide treatment strategies, improve the care of women with advanced endometriosis and infertility, and potentially reduce healthcare costs by identifying the most effective pathway to achieving pregnancy.

DETAILED DESCRIPTION:
WHY THIS TRIAL IS NEEDED

BACKGROUND

Endometriosis Endometriosis is a prevalent condition affecting 10% of female population of reproductive age, leading to pain and sub-fertility. An earlier systematic literature reviews and meta-analysis suggests that women with advanced endometriosis (revised American Society for Reproductive Medicine classification of endometriosis (rASRM) stage III-IV) have a lower likelihood of achieving clinical pregnancy/live birth compared to women without endometriosis, while this difference has not been observed for mild disease (stage I-II).

Gynaecological Ultrasound and staging The prevalence of endometrioma and deep endometriosis found through systematic transvaginal ultrasound on women referred for ART treatment in Sweden has been estimated at 21.8%. Additionally, 75.8% of those with endometriosis were unaware of their condition prior to diagnosis. In recent years, two staging systems, namely the American Association of Gynecologic Laparoscopists (AAGL) Endometriosis classification and #ENZIAN have gained prominence owing to their accuracy when juxtaposed with surgical findings.

Surgical Treatment Women with endometriosis seem to experience pain relief after bowel surgery due to endometriosis. Consensus from the European Society of Human Reproduction and Embryology (ESHRE) indicates that surgery can be performed prior to treatment with assisted reproductive technologies (ART). Additionally, the number of spontaneous pregnancies is high after surgery on patients with deep endometriosis. Furthermore, in patients with endometriosis stage I-II or in infertile patients with endometriomas, surgery can in some cases be considered to improve fertility. However, the risk of severe complications in patients undergoing rectal surgery is up to 10% including anastomosis leakage and fistulas.

Fertility treatment An earlier meta-analysis found that the number of oocytes and fertilization rates are lower in women with endometriosis as compared to those without, although not necessarily impacting the live birth rate. Still, some previous studies have shown lower likelihood of live birth and pregnancy after in vitro fertilisation (IVF) in women with endometriosis compared to women with unexplained or tubal infertility. Even though there is some controversy when it comes to the evidence of association between endometriosis and adverse reproductive outcome after IVF, there is biological plausibility for this type of association, especially in women with advanced endometriosis (chronic inflammation affecting folliculogenesis, technical difficulties at oocyte retrieval due to endometriomas or adhesions, increased risk of pelvic infection after oocyte pick-up).

RATIONALE FOR STUDY

Only a few comparative retrospective studies on first-line surgery versus first-line ART have been performed, with no available randomised controlled trials (RCTs). In two retrospective register studies, first-line surgery in patients with deep endometriosis (DE) in the anterior compartment or colorectal DE showed improved live birth rates (LBR) and pregnancy rates (PR) compared to first-line ART. An important limitation in the previous studies on patients with endometriosis has been the challenge of staging and characterizing the disease consistently using preoperative imaging techniques. Currently, the decision regarding the choice between surgery and IVF is collaborative and individualised, considering various factors such as the patient's medical and surgical history, presence of pain symptoms, age, results of ovarian reserve testing, and semen analysis. Lack of randomised RCTs or at least robust prospective cohort studies comparing these two approaches is noteworthy. Hence, there is an obvious need for a randomised controlled trial to address the impact of surgery prior to ART on the reproductive outcomes in women with endometriosis AAGL stage III-IV, to help patients and health-care workers with decision-making, with the overall aim to improve patient-outcomes.

STUDY OBJECTIVES

HYPOTHESIS First line surgery (prior to ART treatment) in women with endometriosis AAGL stage III-IV will result in improved cumulative live birth rate (CLBR) as compared to first line ART.

PRIMARY OBJECTIVE To assess whether surgery conducted prior to ART treatments in women with endometriosis AAGL stage III-IV increases chances of CLBR as compared to first line ART.

SECONDARY OBJECTIVES

To evaluate whether surgery prior to ART treatments in women with endometriosis AAGL stage III-IV will result in:

* improved cumulative pregnancy rate (CPR) and lower miscarriage rate as compared to first line ART.
* shorter time to live birth or pregnancy as compared to first line ART.
* better reproductive outcomes per IVF cycle and a lower rate of recurrent implantation failure (RIF).
* lower rate of infections after oocyte pick-up requiring treatment with antibiotics as compared to first line ART.
* higher Quality of life and less pain measured with Endometriosis Health Profile (EHP-30) and Numeric Rating Scale (NRS) before ART, i) at the time of oocyte retrieval, ii) two months after ART and iii) at the three-year follow-up visit as compared to first line ART.
* reduced pregnancy and delivery complications, as well as fewer complications within 8 weeks postpartum.

To explore whether surgery prior to ART treatments in women with endometriosis AAGL stage III-IV will be cost effective compared with first line ART.

To investigate whether serum progesterone level on the day of frozen embryotransfer in hormone replacement cycles in patients with severe endometriosis is associated with reproductive outcomes (LBR, pregnancy rate, miscarriage rate) and to determine if there is any difference in p-progesterone level between the two different study groups first line ART vs first line surgery in women with endometriosis AAGL stage III-IV.

PRIMARY OUTCOME MEASURE Cumulative live-birth rate within three years from first treatment (surgery or ART treatment).

SECONDARY OUTCOME MEASURES (see below in the protocol)

STUDY ENROLLMENT

SCREENING PROCEDURE AND PARTICIPANT IDENTIFICATION

All women with stage III-IV AAGL endometriosis with infertility referred and/or eligible for surgery and/or ART-treatment such as IVF or ICSI will undergo screening for this trial. The results of this screening will be documented in a screening log. After obtaining oral and written informed consent, patients will be registered and randomised. Registration data will be entered to an electronic Case Report Form (eCRF).

STAGING

At baseline, a specialised transvaginal and abdominal ultrasound examination, supplemented with transabdominal ultrasound if indicated will be performed according to the International Deep Endometriosis Analysis (IDEA) group recommendations to identify endometriosis lesions. Ultrasound and, if needed, magnetic resonance imaging (MRI) findings will be classified using the #ENZIAN and AAGL classification system.

The presence of adenomyosis will also be documented and characterized according to the Morphological Uterus Sonographic Assessment (MUSA) group recommendation. Women with and without suspected adenomyosis will receive the same treatment protocols. Presence of adenomyosis will not influence allocation but will be considered during the discussion of the final analysis of study results.

The use of hormonal treatment for endometriosis, prior to the surgery/ first ART-treatment or between the surgery and ART-treatment, will be documented and considered in the discussion of the outcomes.

RANDOMISATION

After verification of eligibility, signed informed written consent participants will be randomly assigned to either undergo first-line ART or first-line surgery, followed by ART by equal allocation, 1:1. The randomisation procedure will be stratified for participating center (permuted block design). Randomisation will be performed at each site using the web-based instrument Red Cap. All inclusion criteria and no exclusion criteria must be met. One month before first treatment (IVF or surgery), inclusion and exclusion criteria are entered into the randomisation/registration application RedCap. Patients withdrawn from the study after randomisation but before treatment will be substituted by newly enrolled patients. Patients withdrawn from the study after first treatment will not be substituted. Username and password are required to log in; each investigator authorised to register patients has a personal login username and password. If all criteria are met, patients are registered, and the allocated patient number is recorded in the patients' medical file.

There could be some uncertainty surrounding participants' willingness to engage in a Randomised Controlled Trial (RCT) comparing two fundamentally distinct approaches. Therefore, we intend to offer women who fullfill eligibility criteria but decline randomisation. the opportunity to take part in a parallel study - a prospective cohort study, that would provide valuable real-world outcomes of two different approaches to treatment of endometriosis -associated infertility. This parallel study will evaluate identical outcomes to those in the randomised trial. However, instead of random assignment, participation decisions will be made by the patients themselves, resulting in what is commonly referred to as a patient preference trial.

DEFINITION START OF TRIAL

Start of trial will be defined as start of first treatment which will be either surgery or first ART cycle (e.g. start of FSH injections).

DEFINITION END OF TRIAL

The study will end when all patients enrolled in trial have been followed for 3 years after first treatment, withdrawn consent, or are lost to follow-up. Data from study participants that are lost to follow will be included in the final analysis. The trial steering committee may end enrolment at any time if it is deemed that this is in the best interest of the patients.

STUDY TREATMENT

Time from randomization to first treatment (surgery or first ART cycle) should be minimized with a goal of three months and should preferably not exceed six months. Complications due to treatments (IVF or surgery) will be register in the eCRF and treated according to clinical routine at each hospital.

EXPERIMENTAL TREATMENT

First line endometriosis surgery followed by ART such as IVF or ICSI.

STANDARD/CONTROL TREATMENT

First line ART such as IVF or ICSI.

QUALITY ASSURANCE OF SURGERY AND FERTILITY TREATMENT PARTICIPATING CENTERS

All participating surgical centers have been selected by the National Board of Health and Welfare following an application process to perform highly specialised advanced endometriosis surgery at a national level. A quality assessment form including institutional experience with endometriosis surgery and ART, annual volume of benign gynaecological complex cases must be completed. Moreover, surgical variables (e.g. operation time, blood loss) and complications within 30 days after surgery according to Clavien Dindo (22) must be reported . Furthermore, the infrastructure to participate in the trial must be satisfactory. In addition, the institution's ability to perform staging of endometriosis is considered. All ART-clinics authorised to provide publicly funded fertility care report their results continuously to the National Quality Registry for Assisted Reproduction (Q-IVF).

During the study, it is at the discretion of the coordinating investigators and Trial steering committee to close centers with a higher-than-average rate of postoperative major complications or poor quality of surgery or ART, from further accrual, temporarily or irrevocably after consultation with the Data Safety Monitoring Board.

PARTICIPATING SURGEONS

All included surgeons must be approved by the coordination investigators or/and trial steering committee ensuring adherence to protocol. In the site identification and quality assessment form the participating surgeons experience and annual caseload will be reported for review. It is at the discretion of the coordinating investigators or/and steering committee to select or deselect individual surgeons from participating in the trial. Only surgeons stated in the Quality assessment form are allowed being lead surgeons, amendments during the trial can be made.

Robot-assisted laparoscopic or traditional laparoscopic endometriosis surgery All included surgeons must have a previous experience of at least 20 advanced endometriosis surgeries.

PROSPECTIVE COHORT STUDY

For patients who decline participation in randomization or are excluded after randomization, an option to be included in an observational prospective cohort study will be provided. Participants in this study will adhere to the same study protocol as in the RCT, except for the randomisation itself. Analyses for this cohort will adjust for confounding factors using regression models, as described in the statistical methods section.

LONG-TERM FOLLOW-UP

There will be an opportunity for inclusion in a long-term follow-up, where participants from both the randomised controlled study and the cohort study will be eligible if they consent. In the long-term follow-up, conducted 10 years post-inclusion, we will utilise the unique Swedish personal identification number and gather data after study conclusion on i) infertility treatments from the National Register of ART in Sweden (Q-IVF), ii) live births from the Swedish Medical Birth Register (MFR) and The National Pregnancy Register and iii)number of recurrent endometriosis surgeries from Gynop.

P-PROGESTERONE ON THE DAY OF TRANSFER OF THE CRYOPRESERVED EMBRYO IN HORMONE REPLACEMENT THERAPY-CYCLES

Patients suffering of endometriosis may differ in their response to exogenous progesterone when undergoing frozen embryo transfer cycles (FET) with standard hormone replacement therapy, HRT. The aim of this sub-study is to investigate possible association between P-progesterone levels on the day of FET in HRT cycles and reproductive outcomes. Primary outcome is live birth rate, secondary outcomes include clinical pregnancy rate and miscarriage rate. Potential difference in P-progesterone levels between the two different study groups (surgery first vs IVF first) will also be investigated.

PATIENT REPORTED OUTCOMES (PROMS)

When evaluating quality of life among women with endometriosis many different scales have been used, mostly of generic character that are not specific to the disease. One of these is 30-item Endometriosis Health Profile (EHP30), a scale that perform well in clinical practice in the routine evaluation of Health-Related Quality of life (HRQoL) The use of EHP30 is recommended by the National Board and Welfare in Sweden, the ASRM and ESHRE. Using EHP-30, a small study has shown an improvement in HRQoL in the follow-up after endometriosis surgery, an effect that may last for up to 6.8 years . Two recent studies show postoperative improvement in HQQoL measured by EHP-30 10 weeks and 3 months after surgery, respectively. Especially women with deep endometriosis (DE) showed a more significant benefit from surgery. However, HRQoL can also be affected by infertility, and in this trial, infertility treatment will be delayed in one arm, thus, HRQoL is an important measurement.

HEALTH ECONOMICS

Health economics will be analyzed both with respect to Swedish conditions and with an international perspective.

DIRECT COSTS To evaluate healthcare costs, the internal accounting and billing systems within hospitals will be utilised to estimate direct costs based on Cost Per Patient (CPP) principles for individual treatments and/or Diagnosis-Related Groups (DRG) for surgery and fertility treatment. We will also obtain CPP and/or DRG-based cost data from the hospitals where the included women receive care in connection with surgery, fertility treatment. We will also obtain CPP and/or DRG-based cost data from the hospitals where the included women receive care in connection with surgery, fertility treatments, pregnancy, childbirth, and postpartum follow-up. In addition, data on employment status at baseline will be collected.

INDIRECT COSTS To assess indirect costs related to the disease, both study arms will be examined with regard to estimating productivity costs, specifically the level of decline in production.

STATISTICAL CONSIDERATIONS

The primary exposure is the randomised allocation (surgery prior to ART vs ART alone). All analyses will follow the intention-to-treat (ITT) principle, meaning participants are analyzed according to their randomised group regardless of adherence. Per-protocol and as-treated analyses will be conducted as sensitivity analyses to assess robustness. An interim analysis at the halfway point is planned to monitor potential adverse effects and ensure the safety of the interventions.

No formal adjustment for multiplicity will be made; the primary endpoint will be tested at a two-sided α=0.05, while secondary endpoints are considered supportive and exploratory. Sensitivity analyses will address protocol deviations, handling of missing data, and robustness to alternative modelling approaches.

DATA ANALYSES

Baseline demographic and patient's characteristics will be summarised by treatment group. Continuous variables will be described with mean, standard deviation, median, interquartile range, minimum and maximum, and categorical variables with counts and percentages.

Primary endpoint The primary endpoint of the study is the Cumulative Live Birth Rate (CLBR), defined as the proportion of participants achieving at least one live birth within three years following the initiation of treatment.

Primary analysis The primary analysis will compare proportions between treatment groups and report the crude relative risk (RR) with 95% confidence intervals. Adjusted analyses will use log-binomial regression (or modified Poisson with robust variance if convergence fails), including pre-specified covariates (age, BMI, AMH, ART type, center). A two-sided α=0.05 will be used.

Exploratory subgroup analyses Exploratory subgroup analyses will be conducted using treatment-by-subgroup interaction terms in regression models. Subgroups of interest include type of ART (IVF vs ICSI), age (<35 vs ≥35 years), ovarian reserve (AMH categories), and surgical characteristics (adnexal surgery yes/no; anterior vs posterior deep endometriosis, KVÅ codes). These analyses are exploratory and not adjusted for multiplicity.

Secondary endpoints

Time-to-Event outcomes Cumulative Live Birth Rate (CLBR) and Cumulative Pregnancy Rate (CPR) will be analysed as time-to-event outcomes, defined as the proportion of participants achieving a live birth or pregnancy within three years following initiation of treatment. Kaplan-Meier curves will be used to display cumulative incidence, and groups will be compared with stratified log-rank tests. Treatment effects will be estimated using Cox proportional hazards models, stratified by center and adjusted for pre-specified covariates. Hazard ratios with 95% confidence intervals will be reported.

Cycle-Specific Outcomes Live birth and pregnancy rates per IVF/ICSI cycle will be analysed using log-binomial regression or modified Poisson regression with robust variance to account for within-patient correlation. Other cycle-specific outcomes (e.g. number of oocytes retrieved, fertilisation rate, embryo transfer characteristics, miscarriage rates) will be summarised descriptively and compared between groups using appropriate regression models.

Quality of Life and Health Status Measures:

EHP-30 (continuous, 0-100 scale): Analysed using a linear mixed-effects model (LMM) with random intercepts for participants. Fixed effects will include treatment group, time, and the treatment×time interaction, adjusting for pre-specified covariates (age, BMI, AMH, center).

EQ-5D (continuous index 0-1): Analysed using the same LMM framework as EHP-30 (random intercepts, treatment, time, treatment×time, pre-specified covariates).

NRS pain (ordinal: mild 1-3, moderate 4-6, severe 7-10): Analysed using a generalised linear mixed model (GLMM) with cumulative logit link (ordinal logistic regression), including random intercepts for participants, fixed effects for treatment, time, and treatment×time, and pre-specified covariates (age, BMI, AMH, center).

Health economics A cost-effectiveness analysis will be conducted from the healthcare perspective. Incremental cost-effectiveness ratios (ICER) will be calculated based on QALYs, and probabilistic sensitivity analyses will be performed to address parameter uncertainty.

Additional analysis

* Exploratory subgroup analyses will not be adjusted for multiplicity.
* Safety outcomes will be summarised descriptively by treatment group (frequency, severity, relation to treatment).
* All available data will be used, including outliers.
* Missing outcome data will be handled under the missing-at-random assumption via maximum likelihood in mixed models; for regression models requiring complete covariates, complete-case analysis will be applied.

Covariates Primary and secondary outcomes will be adjusted for pre-specified covariates (age, BMI, AMH, ART type, center), chosen based on clinical relevance and prior evidence.

POWER CALCULATION AND SAMPLE SIZE

The sample size calculation was based on a two-sample comparison of proportions with a two-sided α=0.05 and 80% power. Based on observational data, the cumulative live birth rate (CLBR) after three IVF cycles was assumed to be 55% in the ART-only group and 71% in the surgery+ART group (relative risk ≈1.29). This yields a required sample size of 142 participants per arm (284 total). Allowing for 20% attrition, the planned total sample size is 350 participants.

The necessary sample size for this study is estimated to 323 patients to accommodate a statistical analysis method. This estimation uses the 'pwr' package in R, specifically employing the power.prop.test method, which is designed to compare two proportions. This method is more aligned with contemporary statistical practices and provides a clear, transparent methodology for determining the required sample size based on expected success rates.

This means inclusion of 29 patients from/each center/year and 15 surgeries/year. In a Swedish study published in 2022 the prevalence of endometriosis in patients referred for ART-treatment was 21.8% and 17.2% of women had DE. In 2021 almost 10 500 IVF cycles were performed in Sweden, while more than 5 500 of those were first-time IVF/ICSI with autologous gametes.

INTERIM ANALYSIS AND STOPPING RULES An independent safety and monitoring board (DSMB) will conduct one interim analysis 1.5 years after the randomisation of the first patient or when when 175 patients have completed surgery or first IVF treatment, whichever occurs first. Because each participant has a three-year follow-up and recruitment will be completed within three years, only a limited proportion of primary outcomes will be available at the interim analysis. The analysis will therefore primarily address recruitment feasibility, participant safety including comparison of complication rates between study centers. The DSMB will monitor adverse events in both arms. For surgery, expected complication rates have been described previously in this protocol (9.9% Clavien-Dindo grade 1-2, 3.3% grade ≥3), while ART carries a different spectrum of risks (e.g. ovarian hyperstimulation, infection, or bleeding). A substantially higher-than-expected complication rate in either arm, major discrepancies between centers or other safety concerns may prompt the DSMB to recommend protocol modifications or early termination.

Recommendations from the DSMB will exclusively be communicated to the Trial Steering Committee.

ETHICAL CONSIDERATIONS

RISK-BENEFIT CONSIDERATION By addressing the research questions, we aim to provide evidence to improve patient outcomes in a population that currently faces challenges in fertility treatment due to endometriosis. The research has the potential to benefit participants by improving their chances of successful conception and live birth rates.

Participants in the study may face several direct risks, including physical risks associated with surgery and assisted reproductive technologies, such as infection, or pre- and postoperative complications. Additionally, there may be psychological risks related to the emotional stress of undergoing medical procedures and the uncertainty of treatment outcomes. Furthermore, there are also risks associated with the collection and storage of sensitive medical data, which must be mitigated through robust data protection measures.

In the long term, the research may contribute to improving the understanding and management of endometriosis-related infertility, thereby potentially benefiting future patients.

INSTITUTIONAL REVIEW BOARD/ETHICS COMMITTEE

The study protocol, patient information, and informed consent are approved by Swedish Ethical Review Authority ( dnr: 2024-04293-01, approved 7th October 2024, Amendment, dnr: 2025-03699-02, approved 17th June 2025). Any significant protocol modifications must be submitted to the relevant Independent Ethics Committee or Institutional Review Board for review and approval before implementation. Upon approval from the appropriate committee or board, the investigator will proceed with implementing such protocol modifications. However, in cases of urgent safety concerns, protocol modifications will be promptly implemented without prior approval.

INFORMED CONSENT AND WITHDRAWAL

Before being enrolled in the study, patients will receive both oral and written information on the study objectives, all treatment procedures, and the anticipated and potential adverse events. They will be informed about the strict confidentiality measures regarding their patient data, ensuring that only their treating physician and authorized study personnel will have access to their medical records. Patients will have the freedom to withdraw their consent for study participation at any time, with or without providing a reason, and this decision will not impact their subsequent treatment options or care.

Written informed consent must be obtained from all participants before they are enrolled in the study. The investigator who provided the written and verbal information should also sign the Informed Consent Form during the same encounter. The signed Informed Consent Form should be retained in the Investigator's File, and a copy should be provided to the study participant.

Participants will consent to the following:

* Participation in the study.
* Regulatory authorities and the sponsor's representatives (e.g., monitor) gaining full access to hospital records.
* The control and collection of data for the study.
* The recording, collection, processing, and storage of data in a database.
* Using of data and images for education, lectures, scientific presentations and publications.

PATIENT PROTECTION AND GOOD CLINICAL PRACTICE

The responsible investigator will ensure that the study is conducted in accordance with the principles outlined in the Declaration of Helsinki and/or relevant Swedish or National laws and regulations, whichever offers the highest level of protection for the patient. Participants will be clearly informed that the data collected in the study will adhere to the General Data Protection Regulation (GDPR) (EU 2016/679), ensuring that no subject participating in the study will be identifiable. Women participating in the study will receive treatment in alignment with the international guidelines on Good Clinical Practice (GCP) as defined by the European Parliament (EG596/200).

SUBJECT IDENTIFICATION

Participating patients will be assigned a study-specific code, comprising a two to six-digit number. This code will be utilised for patient registration in the study database. The woman's social identification number will not be included in the database. The key to decipher the code will be accessible solely to the investigator.

GENDER PERSPECTIVE

Endometriosis is a prevalent condition, yet it is rarely acknowledged as a public health concern, despite its pervasive impact across patients' lifecycles. National guidelines were not issued until 2018, and many women with endometriosis report a lack of awareness and understanding of the disease within society. Diagnostic delays are documented in some studies, indicating that patients can suffer from symptoms of this disease up to ten years before a diagnosis of endometriosis is made and treatment is started.

A Swedish epidemiological study conducted in 2019 revealed that 45% of teenage girls experience frequent school absences due to dysmenorrhea, yet only 7% of these girls were given the advice to seek doctor consultation. Sub-fertility often arises as a consequence of endometriosis. In another Swedish study involving women seeking assistance for fertility issues, 75.8% of patients were unaware of their endometriosis diagnosis upon initial consultation at the reproductive medicine center. This suggests that society commonly perceives menstrual pain as a normal discomfort that women are expected to endure.

SIGNIFICANCE OF STUDY

Clinical significance Endometriosis is a prevalent disease among women with infertility, with negative impact on psychological and physical well-being. The management of infertility in women with severe endometriosis is a subject of ongoing debate, with a lack of robust evidence for optimal treatment strategies. Both surgery and ART-treatments in this population may lead to serious complications and are associated with significant costs to society. To date, there are no results from RCTs evaluating potential benefits of endometriosis surgery prior to ART on subsequent reproductive outcomes. This study has the potential to significantly impact the clinical approach to infertility treatment in women with advance endometriosis. Despite the challenges and the coordinated effort required for this RCT, the results promise to be valuable for the scientific and clinical communities.

Implementation Endometriosis is a very prevalent condition (22 % of infertile women) and this research project will indeed affect many patients, regardless of the results. The research group is presently drafting national guidelines for the treatment of infertility in patients with advanced endometriosis. The findings of this study will be integrated into these guidelines to assist decision-making for women with severe endometriosis and infertility.

Additionally, in a consensus document from the European Society of Human Reproduction and Embryology (ESHRE) on endometriosis, it is noted that there is a dearth of randomized controlled trials regarding surgery prior to assisted reproductive technology.

The results of the study will most probably affect guidelines and care for women with severe endometriosis and infertility. It will possibly also lead to insights how to treat women with less severe endometriosis. Other aspects, such as centralisation of advanced surgery as a concept will also be tested.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 38 years old
* Endometriosis AAGL stage III-IV
* Referred or eligible for ART-treatment such as IVF or ICSI, independent of infertility diagnosis (28) (including sperm donation cycles for social reasons) and/or infertility due to dyspareunia/dysmenorrhea caused by endometriosis
* Body mass index 18-35 kg/m2
* Patients who have signed an approved Informed Consent

Exclusion Criteria:

* Previous surgery for endometriosis except diagnostic laparoscopy.
* Previous IVF/ICSI-cycles (including prior fertility preservation cycles)
* Hemato- and/or hydrosalpinx
* Clear indication for surgery such as ureteral stenosis or intestinal sub-occlusive symptoms
* Suspicion of malignancy
* Submucosal fibroids (The International Federation of Gynecology and Obstetrics (FIGO) 0-1, any size) or intramural fibroids (FIGO 2-5, > 4 cm largest diameter of the largest myoma) (29)
* Uterine malformations (class U1-U6 according to ESHRE/ESGE-classification) (30)
* Patients with contraindications to surgery
* Patients undergoing ART with donated oocytes

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2028-09-22 (Estimated); Study Completion 2031-09-22 (Estimated)

PRIMARY OUTCOMES:
Cumulative live-birth rate (CLBR) | Three years from first treatment (surgery or ART treatment)
  CLBR is defined as any live births from first treatment until end of follow up (three years from first ART treatment or surgery or drop out from the study, whichever comes first).

SECONDARY OUTCOMES:
Cumulative Pregnancy Rate (CPR) | From first treatment (surgery or ART) until three years of follow up
  Cumulative Pregnancy Rate (CPR) is defined as all pregnancies confirmed with ultrasound, from first treatment (surgery or ART) until three years of follow up.
Time to pregnancy and live birth | Time is measured up to three years after first treatment
  Time to pregnancy is defined as time from first treatment (surgery or ART) to first pregnancy confirmed with ultrasound. Time to live birth defined as time from first treatment (surgery or ART) to first livebirth.
Spontaneous Pregnancy Rate | between first treatment and end of follow-up (three years)
  Spontaneous pregnancy rate is defined as any spontaneous pregnancy occurring between first treatment and end of follow-up.
Miscarriage rate and/or extrauterine pregnancies | occurring between first treatment and end of follow-up (three years)
  Miscarriage rate defined as frequency and proportion of spontaneous loss of any clinical and biochemical pregnancy before week 22 and/or extrauterine pregnancy defined as a pregnancy not located in the uterine cavity, occurring between first treatment and end of follow-up.
Number of oocytes per IVF/ICSI cycle | At the day of oocyte retrieval for each IVF/ICSI cycle
  Number of oocytes retrieved (mature and total)
Fertilisation rate | The day after oocyte pick-up in each IVF/ICSI-cycle
  Proportion (%) of mature oocytes that became fertilised
Fresh embryo transfer per IVF/ICSI cycle | At the time of transfer or at the end of embryo culture (up to Day 6), per IVF/ICSI cycle
  Fresh embryo transfer - Yes/ No and if Yes - Day 2, 3, or 5
Blastocysts cryopreserved per cycle | at the end of embryo culture (Day 6 after oocyte pick-up)
  Number of blastocysts cryopreserved
Pregnancy outcomes per embryo transfer (ET) | From ET until delivery (up to 10 months)
  Clinical pregnancy rate (confirmed by ultrasound at 6-8 weeks) Miscarriage rate (up to 20 weeks' gestation) Live birth rate (at delivery, up to 10 months after ET)
Cumulative reproductive outcomes per IVF/ICSI cycle | From the start of each IVF/ICSI cycle until completion of all embryo transfers from that cycle (up to 12 months)
  Cumulative pregnancy rate Cumulative miscarriage rate Cumulative live birth rate
Rate of recurrent implantation failure (RIF), (20) evaluated at the end of the study period | Assessed at the end of the study period ( 3 years after randomisation)
  RIF (recurrent implantation failure) evaluated at the end of the study period. RIF is defined here as no pregnancy after three ETs in women <35 years and four ETs in women 35-39 years old (20).
  P-progesterone will be collected on the day of FET, and the test result will be recorded in the eCRF, as a sub-group analysis. The subgroup analysis includes only HRT-FET cycles in patients with endometriosis AAGL stage III-IV diagnosed by ultrasound and surgery. Endometrial preparation is usually performed by using Progynon (4-6 mg/d) per os with the start on the second or third day of menstruation with a possible addition of transdermal estrogen according to local routine. Cyclogest (400 mg/12 h) or other vaginal progesterone preparation of similar efficacy should be commenced when the endometrium is regarded as appropriate by the treating physician (as a rule 7 mm or thicker). Blastocyst transfer should be scheduled on the sixth day of progesterone supplementation (45).
Infections after oocyte retrieval | From each oocyte retrieval and within 2 following months
  Proportion of women in each study arm that are diagnosed with at least one infection after oocyte retrieval ( i.e. within 2 months post-procedure for each IVF/ICSI ), further classified by treatment required: antibiotics only; readmission; surgical intervention
Quality of life and pain | Within 1 month before first intervention; at oocyte retrieval; 2 months after ART or surgery; and at 3-year follow-up.
  Health related quality of life (HRQoL) and pain will be assessed by questionnaires, Endometriosis Health Profile (EHP-30), EQ5D and Numeric Rating Scale (NRS), completed by study participants preferably as electronical patient reported outcome measures or during the clinic visit (by manually filling in forms, by accessible computer or by mail).
  EHP-30 (0-100, higher = worse) EQ-5D (0-1, higher = better) Numeric Rating Scale (0-10, higher = worse pain)
Peri- and two months postoperative complications classified by Clavien-Dindo and Classic systems | Postoperative complications up to two months after surgery
  Intraoperative complications will be classified by Classic systems (21). Two months postoperative complications will be defined according to the Clavien-Dindo (22) system.
Health care costs | From randomization to end of trial
  Health care costs from randomization to end of trial. Direct costs will be used by assessing internal accounting and billing systems within the hospitals, cost per patient (CPP). We will also measure the quality-adjusted life years (QALYs) gained with the intervention and use this to undertake a cost-utility analysis. The QALY calculations will be based on fertility status measures for trial participants, with valuations of changes in fertility status and quality of life based on the EQ-5D
Obstetrical outcomes and complications | From pregnancy week 22 through 8 weeks postpartum
  Proportion of patients in each study arm experiencing Pregnancy-related complications (premature delivery, preeclampsia, gestational diabetes, placenta disorders ) Delivery-related complication (emergency cesarean, pelvic floor trauma, bleeding, manual placenta removal) Postpartum complications (within 8 weeks of delivery: infections, retained tissue, analgesic use)

OTHER OUTCOMES:
P-progesterone levels on the day of frozen embryo transfer in HRT cycle | On the day of frozen embryo transfer (Day 0 of transfer)
  P-progesterone levels on the day of frozen embryo transfer in HRT cycle. Serum progesterone concentration (ng/mL).
Adenomyosis | From first treatment ART or surgery to end of follow-up (three years)
  The presence of suspected adenomyosis, on ultrasound and/or MRI, will be recorded and described at baseline according to Morphological Uterus Sonographic Assessment (MUSA) (26, 27). The presence of adenomyosis will not affect allocation but will be used at the end of the study in the interpretation of the findings, as a sub-group analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Brunes, MD, PhD, Principal Investigator — Karolinska Institutet; Anna Marklund, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Sodersjukhuset, Stockholm, Stockholm County
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Skåne university hospital, Malmö, Malmo
  - Uppsala University Hospital, Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data that underlie the reported results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months following article publication Ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee. A data-sharing agreement will also be required.
  Contact: malin.brunes@regionstockholm.se

REFERENCES:
- See also: Link to the EndoSOFT study published by the Swedish network for national clinical studies in Obstetrics and Gynecology (SNAKS) — https://www.snaks.se/endo-soft/